CLINICAL TRIAL: NCT00228696
Title: National Wilm's Tumor Study Late Effects
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: national study, local site not responsible for results/analysis
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Howard Katzenstein, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB00024842
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Wilm's Tumor
Keywords: late effects
MeSH Terms: conditions — Wilms Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- screening (No Intervention): this is a screening study and no intervention.
  Interventions: Other: none, screening only

INTERVENTIONS:
Other: none, screening only — Screening protocol with no intervention

SUMMARY:
The Late Effects Study is being conducted in order to answer scientific questions and to serve as a resource for Wilms tumor patients and their families. Patients must have been enrolled on the NWTS-5 protocol in order to be eligible for this study.

DETAILED DESCRIPTION:
The Late Effects Study is being conducted in order to answer scientific questions and to serve as a resource for Wilms tumor patients and their families. Although most people in this study enjoy good health, some may be at risk for certain health conditions. We are collecting information from as many participants as possible in order to determine if they or their offspring are at risk for adverse medical conditions. If there is more than one case of Wilms tumor in a given family, we plan to work with geneticists to try to estimate heritability and recurrence risks.

ELIGIBILITY:
Inclusion Criteria:

Previously enrolled in NWTS 5.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
To determine if survivors from Wilms tumors or their offspring are at risk for adverse medical conditions. | 1 year after closure of study

CONTACTS AND LOCATIONS:
Overall Officials: Howard Katzenstein, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States